CLINICAL TRIAL: NCT05992649
Title: The Effect of Aquatic Physiotherapy on Veterans Suffering From PTSD - a 40-week Pilotproject
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: vandfys (Other)
Collaborators: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Lone Nedergaard, Principal investigator physiotherapist, vandfys
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V24
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Single group study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aquatic physiotherapy treatment in warm water (Experimental): The participant is placed supine in the water, supported by the physiotherapist as well as aqua noodles. The physiotherapist supports and moves the participant in the water and adapts to the participant's reaction.
  Interventions: Other: physical therapy

INTERVENTIONS:
Other: physical therapy — Aquatic physiotherapy in warm water

SUMMARY:
Aquatic physiotherapy in warm water pool (AP) is thought to be a helpful treatment for veterans suffering from post-traumatic stress disorder (PTSD). A 40-week program can provide an opportunity to achieve positive results.

Potentiel effects of AP for veterans with PTSD:

Relaxation and stress reduction, anxiety and mood regulation, body awareness and grounding, strength and flexibility and social interactions and camaraderie.

DETAILED DESCRIPTION:
It is estimated that 5% of all veterans who have been deployed have PTSD. In Denmark the total number of deployments are about 27.000 from 1992 - 2012.

The purpose of the project is to investigate the effect of aquatic physiotherapy treatment and physical training in 34-35 degree centigrade warm water in a 40-week program consisting of:

1. st 8 weeks: 30 minutes treatment once a week.
2. nd 8 weeks: 30 minutes treatment once a week +

60 minutes of combined training and relaxation once a week.

3rd 8 weeks: 60 minutes of combined training and relaxation once a week + an activity of own choice once a week.

4th period 16 weeks: 30 minutes treatment once a week + 60 minutes of combined training and relaxation once a week.

Hypothesis:

Veterans with PTSD will experience a reduction in levels of PTSD symptoms.

Methodical approach:

Design: pilot project with an intervention group of 12 receiving treatment and physical training.

Recruitment:

The participants are recruited from Copenhagen Veteran Home, Høvelte Barracks Veteran Home and Military Psychiatric Outpatient Clinic, Rigshospitalet.

cf. inclusion and exclusion criteria.

No of participants to be recruited: 12

Primary effect measures:

Change of PTSD level from baseline using validated questionnaire PCL-M

Secondary effect measures:

1. Change of sleep disorders from baseline using validated questionnaire Pittsburgh Sleep Quality Index (PSQI).
2. Change of self-perceived levels of depression and anxiety by questionnaire (Hopkins symptoms checklist)
3. Change in self-perceived quality of wellbeing measured by questionnaire (WHO-5) Measurements to be taken before and after 24-weeks intervention

Explorative measures:

Change in functionality/ability with everyday life measured by questionnaire (The questionnaire method for assessing functionality/ability

Ethical considerations:

Participation in warm water treatment is considered without side effects or risks.

Using exercise in warm water is part of general physiotherapeutic practice. The treatment is handled by experienced physiotherapists. The project complies with the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* Veteran and have been diagnosed with PTSD.
* Enjoy being in water.
* Have a desire for treatment and training in warm water.
* Will fill out questionnaires and respond to SMS messages related to treatment.
* Speak, read, and understand Danish fluently.
* Will set goals for future participation in local community activities.
* Have practical means to participate (Wednesday and Friday afternoons).
* Can attend treatment or receive assistance with transportation to treatment at Tuborgvej, 2400 Copenhagen NV.
* Any substance abuse should be under control (self-medication, alcohol, and drugs)

Exclusion Criteria:

* fear of water
* physical condition that hinders movement in water
* Fear of getting water in the ears

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-23 (Actual); Primary Completion 2024-07-04 (Estimated); Study Completion 2024-07-04 (Estimated)

PRIMARY OUTCOMES:
Level of symptoms of PTSD | 40-weeks
  Measured by self reported questionnaire PTSD Checklist for military (PCL-M). The self-report rating scale is 0-4 for each symptom (0 = Not at all, 1 = A little bit, 2 = Moderately, 3 = Quite a bit, 4 = Extremely).
  A total symptom severity score (range = 17-85) can be obtained by summing the scores from each of the 17 items. A score between 17-29 suggests little to no severity. A score between 28-29 suggests some PTSD symptoms.

SECONDARY OUTCOMES:
Quality of sleep | 40-weeks
  Measured by self reported questionnaire Pittsburgh Sleep Quality Index (PSQI). In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Levels of symptoms of depression and anxiety | 40-weeks
  Measured by self reported questionnaire Hopkins symptoms checklist. The scale for each question includes four categories of response ("Not at all," "A little," "Quite a bit," "Extremely," rated 1 to 4, respectively). Two scores are calculated: the total score is the average of all 25 items, while the depression score is the average of the 15 depression items, and the anxiety score is the average of the 10 anxiety items. Higher scores indicate worse level of depression and/or anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Bogh Juhl, Professor, Study Chair — Herlev & Gentofte Hospital
Locations (1):
- Lions kollegiets varmtvandsbassin, Copenhagen, Denmark